CLINICAL TRIAL: NCT05642936
Title: A Randomized Controlled Trial of Meditation and Health Education on Carotid Intima-Media Thickness and Major Adverse Cardiovascular Events in Black Women and Men
Brief Title: RCT of Meditation and Health Education on CIMT and MACE in Black Women and Men
Acronym: SR-CIMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi International University (Other)
Collaborators: College of Medicine, Charles R. Drew University of Medicine and Science (Unknown); Barbara Streisand Women's' Heart Center, Smidt Heart Institute, Cedars-Sinai Medical Center, Los Angeles, California (Unknown)
Responsible Party: Principal Investigator, Robert Schneider, MD, Director and Professor, Institute for Natural Medicine and Prevention, Maharishi International University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL51519B
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This was a randomized controlled community-based clinical trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigators and clinic staff were blinded to treatment assignment, except the project manager who did not collect data from participants. Primary care physicians were blinded to the treatment assignments of their patients. Since participants were necessarily aware of their treatment status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcendental Meditation (Experimental): The TM technique is a simple, natural, effortless mental procedure that is practiced 20 minutes twice a day while sitting comfortably with the eyes closed. During the practice, it is reported that ordinary thinking processes settle down, and a distinctive "wakeful hypometabolic" state characterized by neural coherence and physiological rest is gained. The TM technique was taught in a 7-step course of instruction consisting of six 1.5-2 hour individual and group meetings taught by a certified instructor.
  Interventions: Behavioral: Transcendental Meditation technique
- Health Education (Active Comparator): The control intervention was a cardiovascular health education program designed to match the format of the experimental intervention for instructional time, instructor attention, participant expectancy, social support, and other nonspecific factors. The classroom content was based on standard, published materials. The instructors were professional health educators.
  Interventions: Behavioral: didactic health education control

INTERVENTIONS:
Behavioral: didactic health education control — didactic classroom-based comparison group that follows standard guidelines for diet, exercise and substance use with no stress reduction component
  Other Names: lifestyle modification
  Arms: Health Education
Behavioral: Transcendental Meditation technique — a mental technique derived from the Vedic tradition of ancient India and practiced by anyone for 20 minutes twice a day sitting
  Other Names: TM program
  Arms: Transcendental Meditation

SUMMARY:
This was a randomized, single-blind, controlled, community-based trial comparing the clinical efficacy of the Transcendental Meditation program on carotid intima-media thickness and major adverse cardiovascular events in 197 African American men and women at risk for atherosclerotic CVD. After baseline testing, participants were randomly assigned to either a stress reduction program (Transcendental Meditation) or a standard health education program. Follow up was conducted over one year and 12 years.

DETAILED DESCRIPTION:
This was a randomized, single-blind, controlled, community-based trial comparing the clinical efficacy of the Transcendental Meditation (TM) program carotid intima-media thickness and major adverse cardiovascular events (MACE) in 197 African American men and women at high risk for ASCVD. This trial compared the efficacy of the TM program to health education over one year on cIMT. Eligible participants were randomly allocated to either the TM program or health education (HE). The primary outcome was carotid intima-media thickness (IMT) assessed by B-mode ultrasonography at baseline and 12 months. Secondary outcomes were blood pressure, lipids, lifestyle, psychosocial stress and MACE. Fatal and nonfatal clinical events were assessed over one year, and mortality after 12 years.

ELIGIBILITY:
Inclusion Criteria:

race/ethnicity: African American, self-identified, age: no upper limit, gender: male or female, minimum carotid artery intima medial thickness (IMT) of at least .72 mm for men and .65 mm for women or long-term history of diabetes, myocardial infarction, coronary artery revascularization or coronary angiography indicating at least one vessel with 50% stenosis.

Exclusion Criteria:

myocardial infarction, unstable angina, CABG, percutaneous transluminal coronary angioplasty (PTCA), or stroke within the previous three months, carotid artery endarterectomy, arrhythmia - atrial fibrillation, second or third degree AV block, congestive heart failure - class III or IV or ejection fraction less than 30 %, clinically significant valvular heart disease, clinically significant hepatic or renal failure, major psychiatric disorders, current alcohol or other drug abuse dependency disorder, non-cardiac life-threatening illness, and participating in a formal stress management program

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2000-10 (Actual); Primary Completion 2005-07 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Carotid Intima Medial Thickness (CIMT) | 12 months
  This measure of wall thickness of the carotid artery was assessed by B-mode ultrasonography

SECONDARY OUTCOMES:
blood pressure | baseline, 3 and 12 months
  systolic and diastolic BP technique. The three readings were taken one minute apart and then averaged for that visit.
lipid profile | baseline and 12 months
  blood tests or panel for cholesterol, LDL, HDL, and triglycerides
lifestyle factors | baseline, 3 and 12 months
  diet, exercise and substance use
major adverse cardiovascular events (MACE) - fatal and nonfatal | one year
  adverse clinical events - fatal and non-fatal
major adverse cardiovascular events (MACE) - fatal | 12 years
  deaths

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Schneider, M.D., Principal Investigator — Maharishi International University

IPD SHARING:
Plan to Share IPD: Yes
upon request to the study investigators, an outside researcher may inquire for permission to obtain the IPD (deidentified) on an MS excel and Access databases.
Supporting Information: Study Protocol
Time Frame: once the study is published (i.e., in print)

REFERENCES:
- [Derived] Norris KC, Salerno J, Bairey Merz CN, Kaushik V, Gelleta S, Castillo A, Nidich S, Gaylord-King C, Schneider RH. A randomized controlled trial of meditation and health education on carotid intima-media thickness and major adverse cardiovascular events in Black men and women. Front Med (Lausanne). 2025 Mar 19;12:1513699. doi: 10.3389/fmed.2025.1513699. eCollection 2025. PMID 40177279